CLINICAL TRIAL: NCT04108377
Title: Phosphodiesterase 4 Inhibitor, Roflumilast, Improves Beta Agonist Responsiveness Compared to Placebo in Low T2 Asthma Patients.
Brief Title: Phosphodiesterase 4 Inhibitor, Roflumilast, and the Effects of Inhibition in Severe Asthma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Enrollment stopped secondary to completion of funding
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1406843
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-05

CONDITIONS: Asthma
Keywords: Hyperinsulinemia; Phosphodiesterase 4 Inhibitor
MeSH Terms: conditions — Asthma; Hyperinsulinism | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Roflumilast (Experimental): Roflumilast 500mcg by mouth, once daily, for 70 days (10 weeks).
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator): Placebo by mouth, once daily, for 70 days (10 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Roflumilast — Roflumilast capsule
  Other Names: Daliresp
  Arms: Roflumilast
Drug: Placebo — Sugar pill manufactured to mimic look of Roflumilast capsule
  Other Names: Placebo for Roflumilast
  Arms: Placebo

SUMMARY:
This study evaluates the effects of roflumilast on restoring response β2 adrenoreceptor agonists in low T2, obese asthmatics. One group of participants will receive roflumilast for 3 months, while the other will receive a placebo.

DETAILED DESCRIPTION:
T2 low asthma is common in obese asthmatics. New evidence suggests that hyperinsulinemia and insulin resistance, both common in obesity, are associated with an increased risk of concurrent asthma.

Targeting Phosphodiesterase 4 inhibitors (PDE4) allows for examination of a mechanism potentially linking obesity and asthma as well as identification of readily available and safe options to treat hyperinsulinemic, overweight asthmatics.

It is hypothesized that obesity and hyperinsulinemia contribute to asthma by impairing β2 adrenoreceptor function and that this can be rescued the PDE4 inhibitor, roflumilast.

ELIGIBILITY:
Inclusion Criteria:

* Have a physician diagnosis of asthma.
* Require treatment with moderate to high-dose >2500mcg/day of fluticasone or equivalent, or use of oral steroids

Also two of the following:

* Requirement for additional daily treatment with other controller medication
* Daily Asthma symptoms
* Forced Expiratory Volume / Forced Vital Capacity (FEV1/FVC) < 70% and FEV1< 80% predicted
* ≥1 urgent care visits/year
* ≥3 oral steroid bursts/year
* Near-fatal asthma event.
* Exhaled Nitric oxide (FeNO)<30 ppb
* Peripheral blood eosinophil count < 300 (x10-6/ul)
* Obesity, BMI≥30

Exclusion Criteria:

* Less than 18 years of age
* baseline FEV1 <30% predicted
* pregnant or nursing women
* current smokers or subject with >20 pack year history
* any history of intolerance of, or reaction to, Roflumilast.
* Prisoners
* Patients with liver disease
* Subjects with Hepatic impairment (contraindicated in moderate-to-severe liver impairment: Child-Pugh Score Class B/C) for example.
* Patients with clinically significant psychiatric history (i.e., suicidality, etc.) and psychiatric illness
* Patients using strong CYP 450 enzyme inducers (e.g., rifampicin, phenobarbital, carbamazepine, phenytoin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Change in Beta 2 Agonist response from Baseline | 3 months
  Determine whether β2 receptor responsiveness is improved in response to albuterol in Group 1 (Roflumilast) patients compared to Group 2 (Placebo) patients at the study entry.

SECONDARY OUTCOMES:
Exhaled nitric oxide | 3 months
  Determine where exhaled nitric oxide is lower in Group 1 vs Group 2
Asthma Control Test score | 3 months
  The Asthma Control Test (TM © 2002 by QualityMetric) is a validated instrument to measure symptom control in asthma patients. There are 5 questions each with a score of 1-5 (25 total points). Poor asthma control is considered with a score less than 20 out of 25.
  Determine whether Asthma Control Test score is improved in Group 1 vs Group 2
  Asthma Control TestTM
  1. In the past 4 weeks, how much of the time did your asthma keep you from getting as much done at work, school or at home?
  2. During the past 4 weeks, how often have you had shortness of breath?
  3. During the past 4 weeks, how often did your asthma symptoms (wheezing, coughing, shortness of breath, chest tightness or pain) wake you up at night or earlier than usual in the morning?
  4. In the past 4 weeks, how often have you used your rescue inhaler or nebulizer medication (such as albuterol)?
  5. How would you rate your asthma control during the past 4 weeks?

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Kenyon, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis, Sacramento, California, United States

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/a-study-of-the-experimental-medicine-roflumilast-for-severe-asthma-936481/